CLINICAL TRIAL: NCT02997059
Title: Effect of Fluconazole on the Levels of Anti-Saccharomyces Cerevisiae Antibodies (ASCA) After Surgical Resection for Crohn's Disease. Multicenter, Randomized, and Controlled in Two Parallel Groups Versus Placebo
Brief Title: Effect of Fluconazole on the Levels of ASCA After Surgical Resection for Crohn's Disease.
Acronym: AscaMC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited recourse to intestinal resection due to new management of CD
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006_27; 2008-000717-30 (EudraCT Number); PHRC2006R/1903 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Crohn's Disease Aggravated
Keywords: Crohn disease; Candida; ASCA
MeSH Terms: conditions — Crohn Disease; Torulopsis | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluconazole (Experimental): 200mg per day for 6 months
  Interventions: Drug: Fluconazole
- Placebo (Placebo Comparator): One capsule per day for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluconazole — 200 mg/ day
  Arms: Fluconazole
Other: Placebo
  Arms: Placebo

SUMMARY:
This was prospective study randomized in two controlled parallel groups verum versus placebo. The objectives were to assess the influence of antifungal treatment with Fluconazole (FCZ) on the rate of ASCA and endoscopic recurrence at 6 months. The rational was based on our previous research having established i) a link between intestinal inflammation and the opportunistic fungal pathogen C. albicans -a yeast colonizing the human digestive tract- ii) the demonstration that this yeast species could be at the origin of ASCA, a prominent serological marker of CD. It was therefore hypothesized that the FCZ could lower the rate of ASCA and/or reduce the occurrence of recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn disease patients with a small intestine localisation (ileum or ileocecal)
2. Ileal or ileocecal resection in the month before inclusion (resection of all macroscopic lesions). If resection with temporary stoma, the patient may be included at the time of surgery to restore the continuity
3. Patient with low risk of recurrence according to the following criteria:

   (i) Total length of the resection(s) of the small intestine less than 100 cm (ii) Segmental colectomy leaving in place at least another colonic segment as the rectum
4. Preoperative rate of ASCA> 70 arbitrary units (+/- 10%)
5. Informed consent signed to be involved in the study

Exclusion Criteria:

1. Pregnant women or without adequate contraception
2. Total length of the resection(s) of the small intestine more than 1 meter
3. Subtotal colic resection
4. Preoperative rate of ASCA<63 arbitrary units (+/- 10%)
5. Known hypersensitivity to fluconazole or other azoles
6. Known liver disease or transaminase levels >1.5 the normal rate
7. Patient with renal failure
8. Inability to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-07; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of ASCA | 6 months
  the dosage of ASCA in the serum

SECONDARY OUTCOMES:
Identification of yeast digestive colonization | during 6 months
Quantification of yeast digestive colonization | during 6 months
Endoscopic recurrence : Rutgeerts Score>1 | 6 months
Clinical recurrence : surgery for CD (except for proctological surgery) | 6 months
Appearance or not of a clinical recurrence assessed by Crohn Disease Activity Index (CDAI >=220) | 6 months
Number of patients with adverse events as a measure of safety | during 6 months
  Evaluate the clinical and biological safety of the daily dose of fluconazole in this population

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Desreumaux, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sendid B, Salvetat N, Sarter H, Loridant S, Cunisse C, Francois N, Aijjou R, Gele P, Leroy J, Deplanque D, Jawhara S, Weissmann D, Desreumaux P, Gower-Rousseau C, Colombel JF, Poulain D. A Pilot Clinical Study on Post-Operative Recurrence Provides Biological Clues for a Role of Candida Yeasts and Fluconazole in Crohn's Disease. J Fungi (Basel). 2021 Apr 22;7(5):324. doi: 10.3390/jof7050324. PMID 33922391